CLINICAL TRIAL: NCT00979966
Title: Prospective Randomized Phase-II Trial With Temsirolimus Versus Sunitinib in Previously Untreated Patients With Advanced or Metastatic Non-Clear Cell Renal Carcinoma
Brief Title: Study in Non-Clear Cell Renal Carcinoma (Ncc-RCC) Temsirolimus Versus Sunitinib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Central European Society for Anticancer Drug Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-II-006 / 2009-010143-13
Record Dates: First submitted 2009-09-09; First posted 2009-09-18 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Non-clear Cell Renal Cell Cancer
Keywords: Locally advanced or metastatic non-clear cell renal cell cancer (ncc-RCC)
MeSH Terms: interventions — temsirolimus; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Temsirolimus
  Interventions: Drug: Temsirolimus
- B (Experimental): Sunitinib
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Temsirolimus — 25 mg intravenously, once weekly infusion
  Arms: A
Drug: Sunitinib — 50 mg oral once daily for 4 weeks, followed by 2 weeks rest.
  Arms: B

SUMMARY:
This will be a prospective, open-label, randomized multicenter phase-II study to evaluate progression free survival (PFS) in patients with locally advanced or metastatic non-clear cell renal cell cancer (ncc-RCC) receiving Temsirolimus in comparison to Sunitinib.

In most clinical trials in renal cell carcinoma (RCC), clear cell RCC have been included exclusively. There are only some limited data on the efficacy of Temsirolimus or Sunitinib in ncc-RCC showing interesting response rates for both agents. However, randomized clinical trials in this specific patient population have not yet been performed.

In the proposed study a comparison Temsirolimus and Sunitinib is scheduled in first line therapy of ncc-RCC.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males and females: ≥18 years of age.
2. Locally advanced or metastatic, histological confirmed, non-clear cell RCC of all subtypes. Patients must have advanced non-clear cell of one of the following subtypes: papillary, chromophobe, collecting duct carcinoma (CDC), renal medullary carcinoma (RMC), or unclassified.
3. Patients with measurable disease (at least one uni-dimensionally measurable target lesion by CT-scan or MRI) according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) If prior palliative radiotherapy to metastatic lesions: ≥ 1 measurable lesion that has not been irradiated.
4. PS 0-2 ECOG
5. Signed written informed consent.
6. White blood cell count (WBC) ≥4x10*9/L with neutrophils ≥1.5 x 10*9/L, platelet count ≥100x10*9/L, hemoglobin ≥9 g/dL.]
7. Total bilirubin <2 x upper limit of normal.
8. AST and ALT <2.5 x upper limit of normal, or <5 x upper limit of normal in case of liver metastases.
9. Serum creatinine <2.0 x upper limit of normal.
10. Normal ECG without QT prolongation (QTc < 450msec).
11. Adequate cardiac function (left ventricular ejection fraction > 40% as assessed by ECHO.

Exclusion Criteria:

1. Predominant clear-cell RCC
2. Resectability or other curative options
3. Any investigational drug within the 30 days before inclusion.
4. Prior systemic treatment for their RCC.
5. Known or suspected allergy or hypersensitivity reaction to any of the components of study treatments.
6. Radiotherapy within the last 4 weeks.
7. Pregnancy (absence to be confirmed by beta-hCG test) or lactation period.
8. Men or women of child-bearing potential who are sexually active and unwilling to use a medically acceptable method of contraception during the trial.
9. Clinically symptomatic brain or meningeal metastasis. (known or suspected)
10. Cardiac arrhythmias requiring anti-arrhythmics (excluding beta blockers or digoxin).
11. History of any of the following cardiac events within the past 6 months:

    * myocardial infarction (including severe/unstable angina),
    * coronary/peripheral artery bypass graft,
    * congestive heart failure (CHF),
    * cerebrovascular accident,
    * transient ischemic attack,
    * pulmonary embolism.
12. No hemorrhage ≥ grade 3 within the past 4 weeks
13. Uncontrolled severe hypertension (failure of diastolic blood pressure to fall below 90 mm Hg despite the use of ≥3 anti-hypertensive drugs
14. History of relevant pulmonary hypertension or interstitial lung disease.
15. Acute or sub-acute intestinal occlusion or history of inflammatory bowel disease or chronic diarrhea
16. Previous malignancy (other than renal cancer cancer) in the last 5 years except basal cell cancer of the skin, pre-invasive cancer of the cervix or superficial bladder tumor [Ta, Tis and T1].
17. History of organ allograft
18. Significant disease which, in the investigator's opinion would exclude the patient from the study
19. Patients with seizure and epileptic disorder or other conditions requiring medication (such as phenytoin, carbamazepin, phenobarbital)
20. Patients under strong inducers or inhibitors to CYP Isoenzymes
21. Patients with hypersensitivity to the antihistamine or patients who cannot receive the antihistamine for other medical reasons
22. Patients requiring long-term cortisone therapy
23. Patients requiring oral anticoagulation treatment, such as marcoumar. (Anticoagulation treatment with heparin or low molecular weight heparin [LMWH] is allowed provided that close monitoring is performed).
24. Surgery within at least 2 weeks prior to randomization
25. HIV seropositivity.
26. Abnormal pulmonary function (DLCO < 50%). [Pulmonary function tests need only to be performed if abnormal pulmonary function present in medical history].
27. Poorly controlled diabetes mellitus.
28. Liver cirrhosis, chronic hepatitis
29. Legal incapacity or limited legal capacity
30. Known alcohol or drug abuse.
31. Medical or psychological conditions that would not permit the patient to complete the study or sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-07; Primary Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Time to progression | 7-11 months expected

SECONDARY OUTCOMES:
Objective response | 7-11 months expected
safety assessed using CTCAE v3.0 and safety assessed according to reported SAEs | 8-12 months (treatment duration + 1 months)
one year progression free survival rate (1YPFSR) | 1 year
overall survival (OS) | will be evaluated in 2013

CONTACTS AND LOCATIONS:
Locations (14):
- Germany (14):
  - Charité - Campus Virchow Klinikum, Berlin
  - Charité - Mitte, Berlin
  - Vivantes Klinikum am Urban, Berlin
  - Evangelische Kliniken Bonn gGmbH - Johanniter-Krankenhaus, Bonn
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Essen, Essen
  - Klinikum der J.W. Goethe Universität, Frankfurt
  - Martin-Luther-Universität Halle-Wittenberg, Halle
  - Universitätskrankenhaus Jena, Jena
  - UK-SH Campus Lübeck, Lübeck
  - Klinikum Oldenburg gGmbH, Oldenburg
  - Klinikum Stuttgart, Katharinenhospital, Stuttgart
  - Facharzt für Innere Medizin,, Viersen
  - Kliniken Nordoberpfalz AG - Klinikum Weiden, Weiden

REFERENCES:
- [Derived] Aldin A, Besiroglu B, Adams A, Monsef I, Piechotta V, Tomlinson E, Hornbach C, Dressen N, Goldkuhle M, Maisch P, Dahm P, Heidenreich A, Skoetz N. First-line therapy for adults with advanced renal cell carcinoma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 May 4;5(5):CD013798. doi: 10.1002/14651858.CD013798.pub2. PMID 37146227
- See also: German description on the CESAR homepage — http://www.cesar.or.at/